CLINICAL TRIAL: NCT02916069
Title: The Impact Multi Modal Brain Monitoring on Patient Out Come After Adult Cardiac Surgery
Brief Title: Multi Modal Brain Monitoring and Cardiac Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Dr Mohamed Shaaban Ali, PhD, MD, Associate Professor (Anesthesiology and Critical Care)- College of Medicine-Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: IRB00008715621
Record Dates: First submitted 2016-09-16; First posted 2016-09-27 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Intraoperative Neurophysiological Monitoring
Keywords: Spectroscopy; Transcranial Doppler; Bispectral index; Cardiac surgery
MeSH Terms: interventions — Ultrasonography, Doppler, Transcranial; Consciousness Monitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Multimodal brain monitoring) (Active Comparator): Patients will be monitored with combination of brain monitoring; Nearinfrared Spectroscopy (NIRS), Transcranial Doppler (TCD), and Bispectral index (BIS). Interference will be done to optimize the medical condition based on such monitors.
  Interventions: Device: Nearinfrared Spectroscopy (NIRS); Device: Transcranial Doppler (TCD); Device: Bispectral index (BIS)
- Group 2 (No Intervention): Patients will be monitored without any interference based on such monitors

INTERVENTIONS:
Device: Nearinfrared Spectroscopy (NIRS) — Patients will be monitored and interference will be done to optimize the medical condition based on such monitor
  Arms: Group 1 (Multimodal brain monitoring)
Device: Transcranial Doppler (TCD) — Patients will be monitored and interference will be done to optimize the medical condition based on such monitor
  Arms: Group 1 (Multimodal brain monitoring)
Device: Bispectral index (BIS) — Patients will be monitored and interference will be done to optimize the medical condition based on such monitor
  Arms: Group 1 (Multimodal brain monitoring)

SUMMARY:
Multimodal brain monitoring is feasible and can be used in formulating therapeutic strategies during cardiac surgery. Such monitoring may help to improve patient outcome and to reduce costs after cardiac surgery with CPB.

DETAILED DESCRIPTION:
The aim of this study is to use a combination of brain monitoring {Nearinfrared Spectroscopy (NIRS), Transcranial Doppler (TCD), bispectral index (BIS)} to formulate therapeutic strategies based on these monitors and to evaluate the impact on patient outcome.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery with cardiopulmonary bypass
* Valve replacement
* Coronary artery bypass

Exclusion Criteria:

* Emergency surgery
* Hepatic
* Renal impairment
* Diabetes Mellitus

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-03 (Estimated); Study Completion 2018-05 (Estimated)

PRIMARY OUTCOMES:
S100 protein | up to 24 hours
  S100 protein (marker of brain injury)

SECONDARY OUTCOMES:
Mini-mental state examination | up to 30 days after surgery
Western perioperative neurological scale | up to 30 days after surgery
Major neurological out come as stoke | up to 30 days after surgery
Duration of mechanical ventilation | up to 30 days after surgery
Hospital stay | up to 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Ali, PhD. MD, Principal Investigator — associate professor of anesthesia and critical care
Locations (1):
- Faculty of medicine Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided